CLINICAL TRIAL: NCT01794858
Title: Therapeutic Hypothermia for Severe Acute Pancreatitis: A Clinical Model for "Suspended Inflammation"
Brief Title: Therapeutic Hypothermia for Severe Acute Pancreatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S12-00828
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Hypothermia (Experimental): Primary - Organ specific outcome at 28 days Logistic Organ Dysfunction Score (LOD) will be compared before and after TH. Change in LOD will reflect LOD day 4 minus LOD day 1 (Ehrmann, Can J Anesth 2006).
  Secondary
  * Lab values: D-Dimer, IL-6, CRP
  * APACHE II Scores Day 1 and after TH (day 4)
  * Length of stay in the ICU and hospital
  * Prevalence of infections
  * 28-day mortality
  * Hypothermia-related side effects: cardiac arrhythmia, electrolyte balance, hyperglycemia, bleeding, acute pancreatitis
  Interventions: Other: Therapeutic Hypothermia

INTERVENTIONS:
Other: Therapeutic Hypothermia — Will receive medically-necessitated ventilator support under ICU monitoring with core temperatures ≥36°C and severe acute pancreatitis defined as either a Ranson Score ≥7, a CT indicating ≥50% pancreatic necrosis, or a significant deterioration in clinical status including dysfunction of two or more organ systems. All patients will receive current standard management for severe acute pancreatitis and a standardized protocol for application of therapeutic hypothermia and rewarming. Our primary endpoints are organ-specific cardiovascular, respiratory, hematological, renal, and metabolic dysfunction as measured at 28 days. Logistic Organ Dysfunction Scores will be compared before and after therapeutic hypothermia, establishing day 4 versus day 1 changes in LOD.

SUMMARY:
Background: Acute pancreatitis is characterized by a high mortality rate (10%-15%), and a remarkably unpredictable clinical course. Approximately 50% of deaths in acute pancreatitis occur early-within the first 14 days-and early mortality is attributable to sequelae of a severe systemic inflammatory response syndrome (SIRS), which is associated with multi-organ dysfunction syndrome (MODS) that can escalate to renal failure, respiratory failure, and death. Significant improvements in acute pancreatitis mortality will demand innovative approaches to counteract early organ failure. A series of destructive cellular processes begins within minutes of initial pancreatic injury, and the ensuing inflammatory cascade is compounded by disease sequelae including edema, ischemia, and tissue necrosis. Early interventions to reduce inflammation within the first 36 hours have been shown to have significant effects in minimizing progressive organ dysfunction.

Hypothermia is clinically employed to combat cellular injury and systemic responses following ischemia-reperfusion, and is been studied as a mechanism of acute inflammatory inhibition in processes including cardiogenic shock, lung injury, local intestinal injury, and reperfusion injuries to the lung, liver, and endothelium. In numerous studies, effective immunomodulations have been observed including reduction of pro-inflammatory cytokines (TNF-α, IL-6), stimulation of anti-inflammatory cytokines (IL-10), inhibition of pro-apoptotic JNK signaling, reduction of systemic oxidative stress, and inhibition of neutrophils, monocytes, and monocyte-derived macrophages. Most saliently, in the caerulein model of murine acute pancreatitis, therapeutic hypothermia has been shown to reduce serum IL-1, IL-6, and TNF-α, increased serum IL-10, decrease serum amylase and lipase, lower the histological grade of pancreatic injury as compared to normothermic mice, and significant survival benefit. Although therapeutic hypothermia is actively employed in the treatment of traumatic brain injury, neonatal asphyxia, spinal cord injury, and cardiac arrest, no studies have yet been made of its application to acute pancreatitis.

Hypothesis: Patients treated with therapeutic hypothermia (32-34°C) will sustain reduced organ-specific injury in acute pancreatitis.

Proposal: In a Phase IIa pilot clinical trial, we will examine the effects of therapeutic hypothermia on organ-specific outcomes during the early stage of acute pancreatitis. We will recruit five patients aged 18 to 80 receiving medically-necessitated ventilator support under ICU monitoring with core temperatures ≥36°C and severe acute pancreatitis defined as either a Ranson Score ≥7, a CT indicating ≥50% pancreatic necrosis, or a significant deterioration in clinical status including dysfunction of two or more organ systems (defined by ACCP/SCCM Organ Failure Guidelines, Chest 2009). All patients will receive current standard management for severe acute pancreatitis and a standardized protocol for application of therapeutic hypothermia and rewarming. Our primary endpoints are organ-specific cardiovascular, respiratory, hematological, renal, and metabolic dysfunction as measured at 28 days. Logistic Organ Dysfunction Scores (LOD) will be compared before and after therapeutic hypothermia, establishing day 4 versus day 1 changes in LOD. Secondary endpoints include D-dimer, IL-6, C-reactive protein, APACHE II scores on day 1 and day 4, inpatient and ICU length-of-stay, infection, mortality, and hypothermia-associated side effects including cardiac arrhythmia, electrolyte imbalance, hyperglycemia, major bleeding, and acute pancreatitis. We believe that such a study will supply preliminary answers to our chief research questions: does therapeutic hypothermia reduce morbidity as assessed by organ-specific outcomes, does therapeutic hypothermia attenuate the steep rise in inflammation observed in severe acute pancreatitis, and does therapeutic hypothermia shorten the clinical course for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80
2. Intubation with mechanical ventilatory support as medically necessary

2) Cooling device or technique available for >36 hours 3) Core temperature ≥36°C 4) SAP either by:

* Ranson Score of > 7
* CT with pancreatic necrosis greater than 50%
* Significant deterioration of clinical status-dysfunction of 2 or more organ systems (defined by ACCP/SCCM Organ Failure guidelines Chest 2009) 5) ICU monitoring medically necessary

Exclusion Criteria:

1. Patient already receiving therapeutic hypothermia treatment
2. Unlikely to survive for the next 24 hours in the opinion of the ICU Consultant or Surgical Consultant treating the patient
3. Temperature ≤34°C at hospital admission
4. Pregnancy (all female patients of child bearing age who meet the inclusion criteria will undergo a urine pregnancy test).
5. History of Cryoglobulinemia
6. No need for ICU monitoring

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Organ specific outcome | 28 days
  Cardiovascular system dysfunction-either of the following:
  Respiratory dysfunction-either of the following:
  Hematological dysfunction-either of the following:
  Renal dysfunction:
  Metabolic dysfunction: unexplained metabolic acidosis, which was defined as:
  Logistic Organ Dysfunction Score (LOD) will be compared before and after TH. Change in LOD will reflect LOD day 4 minus LOD day 1 (Ehrmann, Can J Anesth 2006).

SECONDARY OUTCOMES:
Treatment Effects | 28 Day Mortality
  * Lab values: D-Dimer, IL-6, CRP
  * APACHE II Scores Day 1 and after TH (day 4)
  * Length of stay in the ICU and hospital
  * Prevalence of infections
  * 28-day mortality
  * Hypothermia-related side effects: cardiac arrhythmia, electrolyte balance, hyperglycemia, bleeding, acute pancreatitis

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Medical Center, New York, New York, United States